CLINICAL TRIAL: NCT01776333
Title: Video Images of Disease for Ethical Outcomes
Brief Title: A Randomized Controlled Trial of a Video Decision Aid in the ICU
Acronym: VIDEO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Angelo E. Volandes, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010-P-001820; 2010-P-001820 (Other: MGH)
Record Dates: First submitted 2013-01-22; First posted 2013-01-28 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Respiratory Failure; Cardiac Event
Keywords: ICU
MeSH Terms: conditions — Respiratory Insufficiency; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual care (No Intervention)
- video arm (Experimental): video decision aid intervention
  Interventions: Behavioral: video decision aid

INTERVENTIONS:
Behavioral: video decision aid
  Arms: video arm

SUMMARY:
Randomized Controlled Trial of a Video Decision Aid in the ICU in surrogates of admitted patients.

ELIGIBILITY:
Inclusion Criteria:

- Age 65 or older Patient does not have the capacity to make decisions Patient admitted to the ICU with life threatening illness including advanced heart, renal, lung, gastrointestinal and oncologic disease Patient has English speaking representative to make decisions on his/her behalf Patient critically ill and unlikely to survive to hospital discharge

Exclusion Criteria:

- Patients who are imminently dying and admitted to the ICU are excluded Wards if the state

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
preference for goal of care regarding medical interventions (e.g., CPR, intubation, etc.) | at baseline admission to the ICU during family meeting up to one week

SECONDARY OUTCOMES:
level of medical care delivered to patient at time of death or discharge from the ICU | at time of death or discharge from the ICU up to one week
anxiety and depression | anxiety and depression at follow up phone call at 3 months after ICU death or discharge
satisfaction with ICU experience | after 3 months from time of death or discharge from ICU
number of medical interventions during ICU stay | during time period in the ICU up to one week

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Volandes, Principal Investigator — MGH
Locations (3):
- United States (3):
  - Cedars Sinai Medical Center, Los Angeles, California
  - BMC, Boston, Massachusetts
  - MGH, Boston, Massachusetts